CLINICAL TRIAL: NCT00023140
Title: Collaborative Study of 1,3 Butadiene Biomarkers
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9401-CP-001
Record Dates: First submitted 2001-08-22; First posted 2001-08-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: biomarkers; exposure; adducts; metabolites; butadiene
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Butadiene is a suspect human carcinogen to which most people are exposed daily. Exposures are difficult to measure by air sampling. This study examines the relationship between air levels and several biomarkers of exposure. Biomarkers are substances analyzed in human tissues or waste products. Adducts are materials formed when a chemical reacts with a biological material. In this study we are looking at biomarkers in the blood: hemoglobin and DNA adducts, and urinary metabolites. If a strong relationship is found then the amounts of biomarkers in a person's blood or urine can tell us how much they have been exposed. The tests are being conducted on petrochemical workers who have a wide range of exposures to butadiene. An international group of investigators is conducting the study.

ELIGIBILITY:
Healthy adults without metabolic disorders

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1999-07; Primary Completion 2002-05 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Harvard School of Public Health, Boston, Massachusetts, United States
- National Chung Kung University, Tainan, Taiwan